CLINICAL TRIAL: NCT00657761
Title: Effect of Enfuvirtide on Lipid and Glucose Metabolism and Mitochondrial Function in Healthy Volunteers
Brief Title: Metabolic Effects of Enfuvirtide in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Jose M Gatell, Hospital Clinic, Barcelona
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: ENF/01FD-05/UF1; EudraCT #: 2005-002018-39
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2008-04-14 (Estimated); Status verified 2008-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Enfuvirtide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Saline solution 0.9% sc/12h for 7 days
  Interventions: Drug: Placebo
- Enfuvirtide (Experimental): Enfuvirtide 90 mg/12h sc for 7 days
  Interventions: Drug: Enfuvirtide

INTERVENTIONS:
Drug: Enfuvirtide — 90 mg/12h sc for 7 days
  Arms: Enfuvirtide
Drug: Placebo — 0.9% saline solution/12h sc for 7 days
  Arms: Placebo

SUMMARY:
The metabolic effects of T-20 are not completely known, since the drug is used in combination with other antiretroviral agents. A short-term study in healthy volunteers, with a double-blind crossover design vs. placebo will illustrate if there may be some direct metabolic effects without the influence of HIV infection and the concurrent use of other drugs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males
* BMI between 19-24.9 kg/m2
* No active concomitant clinical conditions
* Negative HIV, HBV and HCV serologies
* Negative abuse drug urine test

Exclusion Criteria:

* Prior psychiatric illness
* Prior dyslipemia
* Alcohol consumption > 30g/day
* Caffeine consumption > 5 units/day
* Current smoker
* Known drug allergies
* Participation in other drug trials in the previous 3 months
* No medications in the previous 30 days

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2005-09; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Change in fasting plasma total cholesterol | 6 weeks

SECONDARY OUTCOMES:
Changes in LDL- and HDL- cholesterol, triglycerides, oral glucose tolerance test, lactate and mt-DNA | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Neus Riba, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic, Barcelona, Barcelona, Spain